CLINICAL TRIAL: NCT06950463
Title: EFFECT OF CIRCUIT TRAINING ON BONE MINERAL DENSITY IN POST MENOPAUSAL PERIOD
Acronym: CWT and BMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Lotfy Ahmed El-Shater, Physiotherapist, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFFECT OF CIRCUIT TRAINING
Record Dates: First submitted 2025-04-17; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Post Menopausal; Osteoporosis
Keywords: CIRCUIT TRAINING, BONE MINERAL DENSITY, POST MENOPAUSAL PERIOD
MeSH Terms: conditions — Osteoporosis | interventions — WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Intervention Model Description: All patients will be divided randomly into two equal groups (A & B):
  Group A (control group):
  It will be consisted of twenty two post menopausal women who will receive daily dosage of vitamin D3 supplement (600 IU/day) (Schleicher et al., 2016), for 6 weeks as prescribed by the gynecologist, in addition to general advices.
  Group B (Study group):
  It will be consisted of twenty two post menopausal women who will receive the same prescribed program of group (A) in addition to circuit weight training , 50 to 60 minutes/session ,3 sessions per week, for 6 weeks in total. .
  All post menopausal women in both groups (A&B) will be given a full explanation of the study protocol and consent form will be signed by each woman before participating in the study (Appendix I).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients will be divided randomly into two equal groups (A & B): Group A (control group) (Experimental): All patients will be divided randomly into two equal groups (A & B):
  Group A (control group):
  It will be consisted of twenty two post menopausal women who will receive daily dosage of vitamin D3 supplement (600 IU/day) (Schleicher et al., 2016), for 6 weeks as prescribed by the gynecologist, in addition to general advices.
  Group B (Study group):
  It will be consisted of twenty two post menopausal women who will receive the same prescribed program of group (A) in addition to circuit weight training , 50 to 60 minutes/session ,3 sessions per week, for 6 weeks in total. .
  All post menopausal women in both groups (A&B) will be given a full explanation of the study protocol and consent form will be signed by each woman before participating in the study.
  Interventions: Other: Group A (control group): It will be consisted of twenty two post menopausal women who will receive daily dosage of vitamin D3 supplement (600 IU/day) (Schleicher et al., 2016), for 6 week; Device: 1-Dumbbells (set B08Z7SY6SP ,Gymbit , made in China) :They will be used for the treatment procedures of circuit training for all postmenopausal women in group B. Its surface is coated with vinyl fo

INTERVENTIONS:
Other: Group A (control group): It will be consisted of twenty two post menopausal women who will receive daily dosage of vitamin D3 supplement (600 IU/day) (Schleicher et al., 2016), for 6 week — 1-Dumbbells (set B08Z7SY6SP ,Gymbit , made in China) :They will be used for the treatment procedures of circuit training for all postmenopausal women in group B. Its surface is coated with vinyl for scratch resistance and to provide them with a firm grip, even if their hands are sweaty. This dumbbell set consists of two dumbbells weighing 2 kg each, with dimensions of 21.7 x 15.7 x 8.5 cm; 4 kg.
Device: 1-Dumbbells (set B08Z7SY6SP ,Gymbit , made in China) :They will be used for the treatment procedures of circuit training for all postmenopausal women in group B. Its surface is coated with vinyl fo — 1-Dumbbells (set B08Z7SY6SP ,Gymbit , made in China) :They will be used for the treatment procedures of circuit training for all postmenopausal women in group B. Its surface is coated with vinyl for scratch resistance and to provide them with a firm grip, even if their hands are sweaty. This dumbbell set consists of two dumbbells weighing 2 kg each, with dimensions of 21.7 x 15.7 x 8.5 cm; 4 kg.

SUMMARY:
This study will be conducted to determine the effect of circuit training on bone mineral density in post menopausal period.

DETAILED DESCRIPTION:
Female aging involves a transition from a reproductive to non-reproductive state associated with hypoestrogenism. This process comprises pre-menopause, menopause, and postmenopausal. Menopause, defined as the permanent cessation of menstruation resulting from the loss of ovarian follicular activity, marks the end of natural female reproductive life. It is preceded by the menopausal transition, which usually begins in the mid-Forty years old.

Menopause ovarian senescence occurs gradually during the fourth and fifth decades of life, leading to menopause. This senescence results in a changing hormonal milieu, with decreases in the levels of estrogens. That decline affects many tissues of the body ad can produce a variety of signs and symptoms, including vasomotor symptoms, decreased bone density, changes in mood and energy, loss of pubic hair and changes in the genital tissues, as well as effects on sexual function, that all can negatively affect the women's quality of life.

Osteoporosis is a degenerative bone disorder, characterized by thinning and weakening of the bone and a general decrease in bone mass and density. Osteopenia is the previous step before osteoporosis, Menopause negatively affects bone growth. Normally, bones go through a process whereby old bone is replaced with new bone cells, but the body's ability to handle this process changes with age. By around age 35 there is less bone growth. Estrogen is involved in the process of calcium absorption into the bones; thus, due to the drop in estrogen levels, women will experience an accelerated reduction in bone density.

Bone Mineral Density (BMD), is a medical term normally referring to the amount of mineral matter per square centimeter of bones. It is used in clinical medicine as an indirect indicator of osteoporosis and fracture risk (Cole, 2008). Fractures most commonly associated with osteoporosis are those of the hip, the vertebrae, and the wrist. Many clinical guidelines recommend risk factor assessment and measurement of BMD through dual energy X-ray absorptiometry (DEXA) to identify individuals at high risk of fracture.

Strength training is one of the most frequent types of exercise programs applied in order to improve BMD in elderly people. The increased mechanical stress on the bone provided by this type of training has been demonstrated as a causal factor of osteogenesis.

One way to prevent osteopenia and osteoporosis by improving bone metabolism markers is repeated load bearing exercise. A combination of weight-bearing exercise with resistance training is beneficial in people who have suffered bone loss, and this helps to improve functional performance as well as spinal and hip bone density.

Circuit resistance training is an exercise program that has beneficial effects on the cardiovascular system and on improving muscular strength. Such training comprises arrangement, normally 10-15, of safety activities for distinctive body parts. For each one, 12-15 repetitions, utilizing unobtrusive weights (11 and 14 strength of exercises according to Borg scale), are done. Each activity is commonly finished within 30-40 seconds. The subject moves rapidly, starting with one activity, then moving on to the next with a rest of 15-30 seconds between stations. Relying on the level of fitness, the circuit training is repeated one to three times .In this way, circuit resistance training takes around 30 to 40minutes to finish an activity session.

Some studies have demonstrated that the circuit training enhances pulmonary ventilation, O2 consumption, and functional capacity. Furthermore, it improves muscular strength , physical endurance, BMD and improve bone strength. circuit training intervention enhances the bone metabolism by inducing physical stimulation effectively.

Significance of the study:

Insufficient vitamin D levels can also lead to diseases like osteoporosis, osteoarthritis, osteopenia due to bone loss, and increased risk of fractures. The hormone vitamin D is necessary for the absorption of the calcium and also the mineralization of bones which is directly related to BMD. A decrease in vitamin D will result in a decrease in BMD which will directly lead to bone loss and increase the impact of fractures.

Exercise in general, particularly CWT significantly contributes to boosting bone density through mechanical loading, blood hydrogen (PH), and biomechanical modifications to liberate ionized calcium, all of which have a positive impact on bone density. It also improves the health-related physical fitness parameters of cardiovascular fitness, muscular strength, muscular endurance, flexibility, balance, and speed.

However, there were some previous studies investigated how CWT affected older people's general fitness and bone mineral density and found that the circuit training intervention showed positive effects on bone metabolism markers and bone density of old women with osteopenia, being viewed as an effective intervention program applicable in order to prevent and control osteopenia and osteoporosis in line with bone density decrease. But there is lack in the literature review about the effect of circuit training on BMD in post menopausal women .So, This study will be conducted to determine the effects of CWT on bone mineral density, vitamin D level and quality of life of post menopausal women which will be of value and increase the body of knowledge of physical therapists and health care managers in the scientific field.

Delimitations:

This study will be delimited to:

* Forty four postmenopausal women (at least one year after cessation of menstruation).
* Their ages will be ranged from 50 - 60 years old.
* Their body mass index will be less than 30 kg/m2.
* Their T-score of DEXA will be ranged from -1.1 to -2.4.
* All of them must have Vitamin D potential deficiency (insufficiency) from 30 nmol to50nmol.
* All participants must be sedentary life style.

Limitations:

This study will be limited by the following criteria:

* Psychological status of postmenopausal women may affect the study's outcomes.
* Environmental factors may affect the patient's response.
* The daily effort of the participants may affect the result of the study.

Null Hypothesis:

Ho: There is no effect of circuit training on bone mineral density in post menopausal period.

HA: There is an effect of circuit training on bone mineral density in post menopausal period.

Basic assumptions:

It will be assumed that:

* All post menopausal women will answer all questions honestly and will be cooperative during the study procedures.
* They will follow the instructions that will be given to them.
* Clinical methods of evaluation will be reliable and valid.
* All post menopausal women will exert suitable effort as much as possible throughout the treatment procedures.
* All treatment sessions will be conducted at the same level of accuracy.
* Results obtained from the study will be of valuable benefits in women's health field.

ELIGIBILITY:
Inclusion Criteria:

Post menopausal women (at least 12 months after cessation of menstruation. Their ages will range from 50 -60 years old. Their body mass index (BMI) will be less than 30 Kg/m2. All of them have vitamin D potential deficiency (insufficiency) from 30nmol to 50nmol .

Their T-score on DEXA will range from -1.1 to -2.4 indicates osteopenia or low bone density.

They must be able to ambulate independently. All of them must be sedentary life style.

Exclusion Criteria:

All women will be excluded if they have one of the following criteria:

Thyroid, kidney and liver dysfunction. Cardiovascular diseases, severe anemia, uncontrolled diabetes mellitus. Any chest surgery, chronic obstructive pulmonary disease, malignancy. Renal failure, myocardial infarction, myasthenia gravis, hyperthyroidism. Hemorrhage, acute viral disease, acute tuberculosis, mental disorders, or those with pacemakers.

Musculoskeletal disorders or women who received corticosteroids in the last 6 months prior to the study.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 44 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 6 months
  A dual-energy x-ray absorptiometry (Hologic Delphi Dexa Scanner) (DEXA): It will be used to assess the bone mineral density for all women in both groups (A and B) before and after the end of the study program.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient-clinic of Gynecology and Obstetrics in Mashtoul Elsouq Central Hospital, Egypt., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No